CLINICAL TRIAL: NCT04010188
Title: A Registered Observational Cohort Study of Charcot-Marie-Tooth Disease
Brief Title: A Registered Cohort Study on Charcot-Marie-Tooth Disease
Status: Recruiting | Type: Observational
Sponsor: Ning Wang, MD., PhD. (Other)
Responsible Party: Sponsor-Investigator, Ning Wang, MD., PhD., Professor, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: MRCTA,ECFAH of FMU [2019] 192
Record Dates: First submitted 2019-07-04; First posted 2019-07-08 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Charcot-Marie-Tooth Disease
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to analyze the natural history data data from Charcot-Marie-Tooth disease and related disorders in China, to assess the clinical, genetic, epigenetic features of patients with Charcot-Marie-Tooth disease, and to optimize clinical management.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the clinical diagnosis of Charcot-Marie-Tooth disease
* Genetic diagnosis of patients with Charcot-Marie-Tooth disease
* Unrelated healthy controls

Exclusion Criteria:

* Decline to participate.
* Other peripheral neuropathy caused by trauma, immunity and toxicosis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: CMT patients who are diagnosed in the First Affiliated Hospital of Fujian Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2039-12-31 (Estimated); Study Completion 2049-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of Charcot-Marie-Tooth Neuropathy Score (CMTNS) during 6 month | Up to 6 months
  Charcot-Marie-Tooth Neuropathy Score (CMTNS) was first proposed and validated by Shy et al (Neurology, 2005). to provide a reliable measure of impairment in Charcot-Marie-Tooth (CMT). The CMTNS is composed of 9 items evaluating different functions related to the disease: 5 of impairment ('Sensory Symptoms', 'Pin Sensibility', 'Vibration', 'Strength Arms' and 'Strength Legs'), 2 of activity limitations ('Motor Symptoms Arms' and 'Motor Symptoms Legs') and 2 electrophysiological measures. Each item is scored from 0 to 4 and the total sum of the item scores provides a global measure of disease severity, with higher scores indicating worsening function.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Fujian Medical University, Fuzhou, China